CLINICAL TRIAL: NCT05794802
Title: The Effect of Acute Exogenous Oral Ketone Supplementation on Diurnal and Nocturnal Blood Pressure and Glucose Homeostasis
Brief Title: Ketone Monoester and Blood Pressure
Acronym: BHB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-5051
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Blood Pressure
Keywords: ketone monoester; blood pressure; glucose homeostasis; heatlhy adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BHB supplement condition (Experimental)
  Interventions: Dietary Supplement: BHB supplement
- Placebo solution condition (Placebo Comparator)
  Interventions: Other: Placebo solution

INTERVENTIONS:
Dietary Supplement: BHB supplement — Oral consumption of 0.5 g/kg of a BHB supplement (KE4; Ketoneaid®, Falls Church, Virginia, USA)
  Arms: BHB supplement condition
Other: Placebo solution — 80 to 120 ml of a placebo solution, depending on the participant's body weight, with the addition of stevia and bitter agent solution (Bitrex, Scotland, UK) as well as the same flavouring as the ketone supplement drink (provided by Ketoneaid)
  Arms: Placebo solution condition

SUMMARY:
The goal of this clinical trial is to determine the effect of acute consumption of a ketone monoester supplement in healthy male adults.

The main questions it aims to answer are:

* To determine if acute consumption of a ketone monoester supplement modulates diurnal (measured in lab) and nocturnal blood pressure (assessed by ambulatory blood pressure monitoring; ABPM) compared to a taste-matched placebo. The investigators hypothesize that a ketone monoester supplement will acutely decrease systolic and diastolic blood pressure compared to the placebo. The same results are expected for diurnal and nocturnal blood pressure.
* To determine if acute consumption of a ketone monoester supplement improves glucose control measured with continuous glucose monitoring (CGM) following a standardized meal consumed 90 minutes after ingestion of the ketone supplement. The investigators hypothesize that a ketone monoester supplement, consumed 90 minutes before a meal, will decrease the 2-hour postprandial glucose incremental area under the curve (iAUC) and peak glucose compared to a placebo.
* To assess IL-10's ability to inhibit proinflammatory cytokine production (TNF- α and IL-1β) in LPS-stimulated whole blood cultures following the ingestion of β-OHB and placebo. The investigators hypothesize that β-OHB will augment the ability of IL-10 to inhibit TNF-α and IL-1β production compared to placebo.

Using a double-blind placebo-controlled randomized crossover study design, 15 adults will participate in two experimental conditions. Participants will be recruited using a local recruitment database (Nabû), during presentations in community organizations, with posters at the University of Sherbrooke, and from word of mouth.

Following screening, eligible participants will be invited for one baseline and two experimental conditions at the Research Centre on Aging (CdRV). During the baseline visit, the following assessments and tests will be conducted:

* resting heart rate (HR) and blood pressure;
* anthropometry and body composition;
* medical history and questionnaires on physical activity levels, dietary habits and anxiety symptoms;
* explanation of the dietary and physical activity logs;
* installation of accelerometers to control physical activity levels and sedentary behaviors over 10 days and CGM to assess glucose control over the subsequent 10 consecutive days.

During the week following the baseline condition, participants will be invited to the laboratory for their first experimental condition (duration = 240 minutes). Participants will come to the lab in a fasted state (at least 12-hour overnight) to the lab at 8:00 am where following assessments and tests will be conducted:

* resting heart rate (HR) and blood pressure;
* ketone supplement or placebo consumption;
* blood samples and cold pressor test;
* standardized breakfast;
* galvanic skin response;
* visual analog scales assessing gastrointestinal discomfort, hunger and fullness;
* installation of ABPM and explanation of the dietary and physical activity logs.

Forty-eight hours later, participants will complete the same experimental condition with the alternate supplement (ketone or placebo) according to their randomization.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine the effect of acute consumption of a ketone monoester supplement in healthy male adults.

The main questions it aims to answer are:

* To determine if acute consumption of a ketone monoester supplement modulates diurnal (measured in lab) and nocturnal blood pressure (assessed by ambulatory blood pressure monitoring; ABPM) compared to a taste-matched placebo. The investigators hypothesize that a ketone monoester supplement will acutely decrease systolic and diastolic blood pressure compared to the placebo. The same results are expected for diurnal and nocturnal blood pressure.
* To determine if acute consumption of a ketone monoester supplement improves glucose control measured with continuous glucose monitoring (CGM) following a standardized meal consumed 90 minutes after ingestion of the ketone supplement. The investigators hypothesize that a ketone monoester supplement, consumed 90 minutes before a meal, will decrease the 2-hour postprandial glucose incremental area under the curve (iAUC) and peak glucose compared to a placebo.
* To assess IL-10's ability to inhibit proinflammatory cytokine production (TNF- α and IL-1β) in LPS-stimulated whole blood cultures following the ingestion of β-OHB and placebo. The investigators hypothesize that β-OHB will augment the ability of IL-10 to inhibit TNF-α and IL-1β production compared to placebo.

Using a double-blind placebo-controlled randomized crossover study design, 15 adults will participate in two experimental conditions. Participants will be recruited using a local recruitment database (Nabû), during presentations in community organizations, with posters at the University of Sherbrooke and from word of mouth. Following screening, eligible participants will be invited for one baseline and two experimental conditions at the Research Centre on Aging (CdRV). During the baseline visit, the following assessments and tests will be conducted: 1) resting heart rate (HR) and blood pressure; 2) anthropometry and body composition; 3) medical history and questionnaires on physical activity levels, dietary habits and anxiety symptoms; 4) explanation of the dietary and physical activity logs; 5) installation of accelerometers to control physical activity levels and sedentary behaviours over 10 days and CGM to assess glucose control over the subsequent 10 consecutive days. Informed consent will be obtained from all participants involved in the study before participating in any assessments or tests. The participant will then be invited to our lab for two non-consecutive days for the experimental condition (at least 48 hours apart).

The first visit will take place at the CdRV (Sherbrooke, QC) on a Thursday or Friday morning. Once the informed consent has been obtained, a medical history and a physical activity questionnaire (International Physical Activity Questionnaire) will be completed by the participant. Body weight, height, and waist circumference will then be measured using standardized procedures. Body composition will be assessed using Dual Energy X-ray absorptiometry (DXA). A CGM will be installed at the abdominal region by the participant himself with the supervision of an experienced exercise physiologist. To limit compensatory behaviours in response to observed blood glucose levels, CGM will be blinded to participants. Finally, participants will be outfitted with a thigh-worn activPAL4 and a hip-worn ActiGraph wGT3X-BT accelerometer to wear for the following 10 days. Wearing the accelerometers will allow for comparing physical activity levels and sedentary behaviours on the days before and after each condition. To ensure that both accelerometers provide reliable data, standardized tests will be performed in our laboratory during the baseline condition. While wearing the activPAL4 and ActiGraph, participants will walk on the treadmill (Life Fitness, Club Series, FlexDeck®; Rosemont, IL, USA) at 3.0, 5.0 and 7.0 km/h for 6 minutes at each intensity. Participants will also have to be in a seated, recline and lying position for 5 minutes each and perform non-ambulatory tasks (washing dishes - 6 minutes and setting the table - 3 minutes). All participants will wear the Xsens motion system during these tasks to capture movement and inform us of the activity profile for better data analysis.

During the week following the baseline visit, participants will be invited to the CdRV for the first experimental condition (duration = 240 minutes). Participants will come to the lab in a fasted state (at least 12-hour overnight) to the lab at 8:00 am where resting blood pressure will be measured in a standardized manner. HR will be continuously monitored for the duration of the visit in the lab (from 8:00 am to 12:00 pm) using a heart rate monitor (Polar H10, Kempele, Finland). At 8:20 am, blood samples will be collected by a certified research nurse. A total of 35 mL of blood will be collected in EDTA tubes for whole blood culture and CPT sodium heparin tubes for PBMC isolation and subsequent transcriptomic analyses. Capillary β-OHB levels will be measured using the Abbot Freestyle Precision Neo® ketone meter before the ingestion of the ketone monoester supplement drink or the taste-matched placebo. At 8:30 am participants will be allowed 2 minutes to consume the oral ketone supplement or placebo drink (liquid form; ~80 - 120 mL depending on to the participant's body weight). β-OHB concentration will then be measured at 30, 60, and 90 minutes after ingestion (~9:00, 9:30, and 10:00 am). Participants will remain seated for 90 minutes following ingestion of the ketone supplement while standardized blood pressure measures will be performed every 20 minutes. At 9:30 am (i.e., 60 minutes after β-OHB ingestion), another blood sample collection will be done (25 mL). Five minutes after the blood sample collection, and right before the blood pressure challenge (i.e., cold pressor test), resting blood pressure and HR will be measured. The cold pressor test will allow the evaluation of the vascular response following an external stressor in a controlled setting, which can occur in everyday life, following the consumption of β-OHB.

Ninety minutes after ketone or placebo ingestion, participants will consume a standardized breakfast consisting of a meal replacement drink, granola bars, and orange juice, which is representative of a realistic mixed meal (MMTT) and provides 490 kcal (68g CHO, 12g FAT, 29g PRO; 55%, 22%, and 23% respectively). Participants will then remain seated for 120 minutes after the MMTT to assess glucose response (CGM) in the postprandial state, and blood pressure will be measured every 20 minutes. Additionally, participants will be asked to complete visual analog scales assessing gastrointestinal (GI) discomfort at -10, 0, 30, 60 and 90 minutes after ketone supplement consumption to monitor for GI distress. Participants will also be asked to complete visual analog scales for hunger and fullness at -10, 0, 60 and 90 minutes after the standardized meal. At 12:00 pm, participants will then be outfitted with the ABPM (IEM PWA Mobil-o-graph; I.E.M. GmbH, Germany) on the non-dominant arm with the appropriate cuff size as suggested by the manufacturer. Participants will also receive instructions on how to fill the logbook, which asks participants to record bedtime hours, physical activity, and sleep quality (assessed via a visual analogue scale). Nutritional intake will be estimated by using the Keenoa app.

Another ketone supplement or placebo drink will be provided to consume directly before going to bed.

Participants will be asked to refrain from structured exercise, alcohol, and caffeine consumption, limit physical activity to their activities of daily living on the day before and during each trial, and replicate their dietary intake 24 hours before and 24 hours after both experimental visits. Furthermore, participants will also be asked to refrain from taking any medications that could affect glucose metabolism or blood pressure and any short-term analgesics (acetaminophen, ibuprofen, etc.). While being conducted in free-living settings, standardizing the experimental conditions as outlined above will allow for controlling any potentially confounding factors between both conditions that could affect our variables of interest and therefore improve measurement rigour.

Forty-eight hours later, participants will complete the same experimental condition with the alternate supplement (ketone or placebo) according to their randomization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male
* 20 to 45 years old

Exclusion Criteria:

* Changes in any type of medication in the last 6 months
* Individuals taking beta-blocker
* Prior history of cardiovascular disease or stroke
* Individuals following a ketogenic diet, low-calorie diet, periodic fasting regimen or consuming ketogenic supplements
* Currently smoking
* Unable to read or communicate in french or english

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure and ambulatory blood pressure | Baseline, before supplements' ingestion, each 20 minutes post-dose and during the subsequent 24 hours
  Resting systolic and diastolic blood pressure (BP) will be measured after 5 minuntes of rest, in a sitting position using an automatic BP monitor (Spot Vital Signs LXi, Welch Allyn Inc., NY, USA). Three BP measurements will be taken interspersed with 1 minute between measurements. If a variation greater than 5 mmHg for BP is observed, a maximum of two more measurements will be taken. During the condition, blood pressure will be measured every 20 minutes. Ambulatory blood pressure will be performed over 24 h using ambulatory blood pressure monitoring (ABPM, IEM PWA Mobil-o-graph; I.E.M. GmbH, Germany). The ABPM will be installed on the non-dominant arm and BP will be measured every 20 minutes after the condition (after 12:00 pm) and every 30 minutes during the night. The nocturnal period will be determined with the participant before every condition.
Effect on glucose homeostasis | Baseline and during the next 10 days
  During the first visit to the CdRV, a continuous glucose monitor (CGM, G6™ sensor, Dexcom Inc., San Diego, CA, USA) will be installed on the arm of the participant, which is to be worn for the subsequent 10 days. During this period, the CGM will collect the following data: blood glucose following ingestion of the ketone supplement (90 minutes), postprandial blood glucose (for 2h following the standardized meal), 24-hour blood glucose, time in range, time spent in hyperglycemia (> 10 mmol/L), hypoglycemia (< 3.8 mmol/L), and mean nighttime blood glucose. For glycemic variability, the following indices will be calculated with Macros in Excel (Easy GV; version 9.0): standard deviation (SD), CV%, and CONGA1 (continuous overall net glycemic action). The CGM will be removed 24 h after the last experimental condition. Raw data will be downloaded from the monitor and analyzed using the Clarity platform (Dexcom Inc., San Diego, CA).

SECONDARY OUTCOMES:
Changes in IL-10 inflammatory profile | 10 minutes pre-dose and 60 minutes post-dose in each condition
  Whole blood cultures will be used to assess IL-10's ability to inhibit proinflammatory cytokines secretion. Briefly, 800 µL of EDTA whole-blood will be diluted 10-fold in Roswell Park Memorial Institute (RPMI) cell culture media. Whole blood will be stimulated with 1 ng/mL of liposaccharide (LPS) in the presence or absence of different IL-10 concentrations (0, 1, 2.5, 5, 10 ng/mL) and incubated for 4 hours at 37°C and 5% CO2. To assess the dose response of β-OHB alone on pro- (TNF-α, IL-1β) and anti-inflammatory (IL-10) cytokines, separate wells containing 10-fold diluted blood will be treated with different β-OHB concentration (1, 2.5, 5 and 10 mmol/L). Unstimulated and LPS only wells will be included to determine the impact of β-OHB ingestion on basal and stimulated cytokine secretion from whole blood. Cytokine concentrations will be determined in culture supernatants using commercially available multiplex kit (Luminex technology).
Changes in transcriptomic analyses of peripheral blood mononuclear cells | 10 minutes pre-dose and 60 minutes post-dose
  As cytokine production is mainly driven by peripheral blood mononuclear cells (PBMC) in whole blood cell culture, peripheral blood collected in CPT heparin tubes (BD sciences) before and 60 minutes after the β-OHB and placebo consumption will be used to isolate PBMC by density gradient centrifugation. Isolated PBMC will be frozen in TRIzol reagent (Invitrogen, Life technology) for a final cell density of 5 x10*6 cells per vial and use for targeted transcriptomic analyses (IL-6, TNF-α, IL-1β and IL-10). Complete blood counts will be performed to account for the daily variability in immune cells count and function with whole blood (EDTA tube) sent to the CIUSSS de l'Estrie - CHUS laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Eléonor Riesco, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No